CLINICAL TRIAL: NCT00358228
Title: Comparison of the Efficacy and Safety of 2 Oral Doses of Rimonabant, 5 mg/Day or 20 mg/Day, Versus Placebo, as an Aid to Smoking Cessation (STRATUS US, EFC4964) - A Randomized, Double-blind, 3-arm, Placebo-controlled, Parallel-group, Fixed-dose, 52-week, Multi-center Study.
Brief Title: Comparison of the Efficacy and Safety of 2 Oral Doses of Rimonabant, 5 mg/Day or 20 mg/Day, Versus Placebo, as an Aid to Smoking Cessation (STRATUS US)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC4964; SR141716
Record Dates: First submitted 2006-07-28; First posted 2006-07-31 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Abstinence
MeSH Terms: conditions — Smoking Cessation | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Rimonabant

SUMMARY:
The primary study objective was to assess the efficacy of 2 fixed doses of rimonabant versus placebo on abstinence from tobacco use in cigarette smokers.

The secondary study objectives were:

* To evaluate the effects of rimonabant on craving and weight;
* To evaluate the clinical and biological safety and tolerability of rimonabant in a population of cigarette tobacco smokers during a 10-week treatment period
* To evaluate the population pharmacokinetics of rimonabant (ie, standard PK evaluation in the population of smokers);
* To observe the percentage of abstinent patients during a 40-week follow-up post treatment period;
* To evaluate quality of life (QOL) and pharmacoeconomics.

ELIGIBILITY:
Inclusion Criteria:

* Smokers smoking at least 10 cigarettes/day (on average) in the 2 months preceding screening visit;
* Motivated to quit smoking (Motivation Scale Score above or equal to 6 on a 10-point scale).

Exclusion Criteria:

* Smoked or consumed more than 3 times within the 3 months immediately preceding the screening visit: non tobacco cigarettes or related products or any form of tobacco product other than cigarettes;
* Current and regular consumption of marijuana (hashish).
* Met current criteria on the MINI International Neuropsychiatric Interview (MINI) for any of the following psychiatric disorders/states: major depressive episode, dysthymia, suicidality, manic episode or hypomanic episode, panic disorder, agoraphobia, social phobia (social anxiety disorder), obsessive compulsive disorder, posttraumatic stress disorder, alcohol dependence or abuse, substance dependence or abuse (excluding nicotine or caffeine), anorexia nervosa, bulimia nervosa, or generalized anxiety disorder;
* Met lifetime criteria on the MINI for manic episode or hypomanic episode, or psychotic disorders;
* Carried a diagnosis of, or suspicion of any cognitive disorder (eg, delirium, dementia, amnestic disorder) or any other psychiatric or developmental disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) that may interfere with his/her ability to understand or complete study related procedures;
* Had a history of severe depression, ie, those who have required hospitalization, or patients with 2 or more recurrent episodes of depression, or a history of multiple suicide attempts;
* Had used, within 3 months before the screening visit:

  * Nicotine replacement of any type for more than 3 days at the maximum prescribed dose, or
  * Behavioral and/or motivational counseling, therapy, support group, or other procedure intended to assist smoking cessation on more than 3 days, or
  * Bupropion (amphebutamone), or
  * Systemic long acting corticosteroids, or
  * Any therapy intended to treat or alleviate depressive symptoms (pharmacologic, somatic, or psychological) for more than 1 week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 787 (Actual)
Dates: Start 2002-09; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Prolonged abstinence from tobacco smoking during the last 4 weeks of treatment (Day 43 to Day 70) as reported by direct inquiry of the patient by the Investigator, and confirmed by exhaled carbon monoxide (CO) levels, and plasma cotinine measurements.

SECONDARY OUTCOMES:
Analysis of mean change from baseline to last evaluation of the total score of QSU.
Brief scale evaluating craving for tobacco cigarettes and relative change in body weight from baseline to last evaluation in patients with BMI lower than 30 kg/m2 at baseline achieving prolonged abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Lowell C. DALE, MD, Principal Investigator — Mayo Clinic 200 First Street SW, Rochester, Minnesota 55905, US
Locations (1):
- Sanofi-Aventis Administrative Office, Malvern, Pennsylvania, United States